CLINICAL TRIAL: NCT04497324
Title: PERUCONPLASMA: Randomized Clinical Trial to Evaluate Safety and Efficacy of the Use of Convalescent Plasma in Hospitalized Patients With COVID-19
Brief Title: PERUCONPLASMA: Evaluating the Use of Convalescent Plasma as Management of COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PER-016-20; 20997 (Registry Identifier: Peruvian Clinical Trial Registry (REPEC))
Record Dates: First submitted 2020-07-31; First posted 2020-08-04 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-03

CONDITIONS: COVID-19
Keywords: COVID-19; Convalescent plasma
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Administration of 1 to 2 units of convalescent plasma (200 ml to 250 ml, each), within 48 hours, plus standard of care.
  Interventions: Biological: Convalescent plasma
- Control group (No Intervention): Standard of care

INTERVENTIONS:
Biological: Convalescent plasma — Administration of 1 to 2 units of convalescent plasma (200 ml to 250 ml, each), within 48 hours, plus standard of care.
  Arms: Experimental group

SUMMARY:
Open label controlled clinical trial to evaluate the safety and efficacy of the use of convalescent plasma in hospitalized patients with COVID-19 infection. This study will have two arms, one arm will receive convalescent plasma plus standard of care, and the other arm will receive standard of care only. Adults older than 18 years old, hospitalized with diagnosis of COVID-19 confirmed by a laboratory test (molecular or serology), with severe or life-threatening disease, will be included to the study after obtaining inform consent by the patient of a direct family member. Participants will be then randomized 1:1 to the experimental and the control groups.

Participants at the experimental group will receive 1 to 2 units of ABO compatible COVID-19 convalescent plasma (200 ml to 250 ml each) within 48 hours, in addition to the standard of care. Participants at the control group will receive standard of care. Safety of convalescent plasma administration will be evaluated, as well as other indicators of clinical efficacy.

DETAILED DESCRIPTION:
The study protocol can be found in:

https://trialsjournal.biomedcentral.com/articles/10.1186/s13063-021-05189-6

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized 18 years old or older patient with COVID-19 disease, confirmed by a molecular test or a serologic test, along with a typical COVID-19 clinical presentation.
* Severe or critical disease caused by COVID-19 Severe disease is defined as 2 or more of the following criteria:

  * Respiratory frequency >22
  * O2 saturation ≤93%
  * PaO2 50mmHg
  * PaO2/FiO2 <300
* Or critical disease with one or more of the following criteria:

  * Respiratory insufficiency with requirement of mechanical ventilation within the last 72hours
  * Shock
* Inform consent signed by patient or direct family member.

Exclusion Criteria:

* Contraindication for transfusion (history of TRALI or TACO, history of anaphylaxis to blood components
* Multiorgan failure, defined by a SOFA score of >5
* hemodynamically unstable, with mean arterial pressure <60 mmHg, refractory to vasopressors use
* Uncontrolled concomitant infection
* Disseminated intravascular coagulation
* Myocardial infarction
* Acute coronary disease
* Patient on dialysis
* Intracranial bleeding active within the last 7 days
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-04-17 (Actual); Study Completion 2021-04-17 (Actual)

PRIMARY OUTCOMES:
Transfusion-related Serious Adverse Events | 14 days after randomization
  Incidence of transfusion-related Serious Adverse Events, according to the Hemovigilance Module Surveillance Protocol v2.5.2

SECONDARY OUTCOMES:
All-cause in-hospital mortality | 30 days after randomization
  Death during hospitalization within the first 30 days after enrollment
Length of hospital stay | 30 days after randomization or until hospital discharge, whatever comes first
  Number of days from date of enrollment to date of discharge
Length of ICU stay | 30 days after randomization or until hospital discharge, whatever comes first
  Number of days from date of admission to the ICU to date of discharge from ICU
Need of invasive mechanical ventilation | 30 days after randomization or until hospital discharge, whatever comes first
  Requirement of invasive mechanical ventilation (Yes/No). Evaluated only for those participants that were on non-invasive ventilatory support at time of randomization
Duration of mechanical ventilation | 30 days after randomization or until hospital discharge, whatever comes first
  Number of days from date of intubation to date of successful extubation
Clinical Improvement at 14 days | At 3, 14 and 30 days after randomization
  Improvement of 2 or more points in the WHO progression scale

CONTACTS AND LOCATIONS:
Overall Officials: Fiorella Krapp Lopez, MD, MSc, Principal Investigator — Universidad Peruana Cayetano Heredia; Patricia Garcia Funegra, MD, MSc, Principal Investigator — Universidad Peruana Cayetano Heredia
Locations (2):
- Peru (2):
  - Hospital Cayetano Heredia, Lima
  - Hospital Nacional Hipolito Unanue, Lima

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Soto A, Krapp F, Vargas A, Cabrejos L, Argumanis E, Garcia PL, Altamirano K, Montes M, Chacon-Uscamaita PR, Garcia PJ. Randomized clinical trial to evaluate safety and efficacy of convalescent plasma use among hospitalized patients with COVID-19 (PERUCONPLASMA): a structured summary of a study protocol for a randomized controlled trial. Trials. 2021 May 17;22(1):342. doi: 10.1186/s13063-021-05189-6. PMID 34001174